CLINICAL TRIAL: NCT05697211
Title: A Pilot Study to Explore Safety, Tolerability and Efficacy of ORal IrON Supplementation with Ferric Maltol in Treating Iron Deficiency and Anaemia in Patients with Heart Failure
Brief Title: ORal IrON Supplementation with Ferric Maltol in Treating Iron Deficiency and Anaemia in Patients with Heart Failure (ORION-HF)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hannover Medical School (Other)
Collaborators: Norgine (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ORION-HF
Record Dates: First submitted 2022-08-18; First posted 2023-01-25 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Heart Failure, Left-sided; Anemia, Iron Deficiency
Keywords: Iron Deficiency
MeSH Terms: conditions — Heart Failure; Anemia, Iron-Deficiency; Iron Deficiencies | interventions — ferric maltol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Feraccru® 30 mg hard capsules (Experimental): Treatment with Feraccru® 30 mg hard capsules (Ferric maltol 30 mg). One capsule twice daily p.o., morning and evening, on an empty stomach
  Interventions: Drug: Ferric maltol 30 mg (Feraccru®)

INTERVENTIONS:
Drug: Ferric maltol 30 mg (Feraccru®) — In this trial Feraccru® 30 mg hard capsules will be used. Each capsule contains 30 mg iron (as ferric maltol), 91.5 mg of lactose, 0.5 mg of Allura Red AC (E129) and 0.3 mg Sunset Yellow FCF (E110) as excipients with known effects.

SUMMARY:
This is an open-label, single arm, multicenter pilot-study to explore the safety, tolerability and efficacy of oral iron supplementation with ferric maltol in treating iron deficiency and anaemia in patients with heart failure.

ELIGIBILITY:
Inclusion Criteria:

1. Men, women*, inter/diverse aged ≥ 18 at day of inclusion
2. Signed written informed consent from patient prior to any study-related procedure and willingness to comply with treatment and follow-up procedures
3. Patients capable of understanding the investigational nature, potential risks and benefits of the clinical trial
4. Patients with chronic heart failure with an Left ventricular ejection fraction (LVEF)<50% (Heart failure with reduced ejection fraction (HFrEF), Heart failure with a mid-range ejection fraction (HFmrEF)) or patients with chronic heart failure with an EF≥50% (HFpEF) and New York Heart Association functional class II-IV
5. 6 min walk distance >50 m
6. Mild-to-moderate anaemia and iron -deficiency as defined by a haemoglobin concentration ≥8 g/dl and <12 g/dl in females or ≥9 g/dl and <13 g/dl in males, and serum ferritin <100 µg/l, or 100-299 µg/l and transferrin saturation <20% at screening
7. *Women without childbearing potential defined as follows:

   * females before menarche (if applicable)
   * at least 6 weeks after surgical sterilization by bilateral tubal ligation or bilateral oophorectomy or
   * hysterectomy or uterine agenesis or
   * ≥ 50 years and in postmenopausal state > 1 year or
   * < 50 years and in postmenopausal state > 1 year with serum Follicle stimulating hormone (FSH) > 40 IU/l and serum estrogen < 30 ng/l or a negative estrogen test, both at screening or

     *Women of childbearing potential:
   * who are practicing sexual abstinence (periodic abstinence and withdrawal are not acceptable) or
   * who have sexual relationships with female partners only and/or with sterile male partners or
   * who are sexually active with fertile male partner, have a negative pregnancy test during screening and agree to use reliable methods of contraception** from the time of screening until end of the clinical trial.

     * The following methods of contraception are acceptable): e.g.

       * progestogen-only oral hormonal contraception, where inhibition of ovulation is not the primary mode of action
       * male or female condom with or without spermicide
       * cap, diaphragm or sponge with spermicide

Exclusion Criteria:

1. Active haematological disorders other than anaemia and/or iron -deficiency
2. Other medical condition that according to the investigator's assessment is causing or contributing to anaemia
3. Active malignancy or currently receiving chemotherapy or radiotherapy
4. Active infectious disease
5. Active bleeding
6. Severe renal insufficiency (glomerular filtration rate (GFR) < 20ml/min or requiring dialysis)
7. Severe liver injury as indicated by serum aminotransferases >3 x upper limit of normal or bilirubin levels >50 µmol/l
8. Ongoing oral or intravenous iron supplementation
9. Concomitant erythropoietin medication
10. Erythropoiesis stimulating agents (ESA), i.v. iron or blood transfusion administered in last 3 months and oral iron (>100 mg/day) in previous 4 weeks
11. Pregnancy or lactation period
12. Subject has received any investigational medication or any investigational devices within 30 days prior to the first dose of study medication or is actively participating in any investigational drug/ devices trial, or is scheduled to receive investigational drug/devices during the course of the study
13. Known or suspected hypersensitivity to any of the active substances or any excipients of the investigational medicinal product
14. Known haemochromatosis or other iron overload syndromes
15. Patients with severe, uncorrected valvular heart disease
16. Clinical evidence of Acute coronary syndrome (ACS), Transient ischaemic attack (TIA) or stroke within the last 30 days
17. Coronary artery bypass graft (CABG), Percutaneous transluminal coronary angioplasty (PTCA), cardiac device implant/resynchronisation therapy or major surgery leading to significant blood loss within last 30 days
18. Planned CABG, PTCA, cardiac device implant/resynchronisation therapy or major surgery
19. Anaemia due to reasons other than iron deficiency (e.g., haemoglobinopathy). Subjects with Vitamin B12 or folic acid deficiency who in the opinion of the Investigator are stable and asymptomatic will be permitted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-02-21 (Actual); Primary Completion 2025-01-08 (Actual); Study Completion 2025-01-08 (Actual)

PRIMARY OUTCOMES:
Change in haemoglobin level from baseline to week 16 | baseline to week 16

SECONDARY OUTCOMES:
Change in serum ferritin from baseline to week 16 | baseline to week 16
Change in transferrin saturation from baseline to week 16 | baseline to week 16
Change in soluble transferrin receptor 1 from baseline to week 16 | baseline to week 16
Change in 6 min walking distance from baseline to week 16 | baseline to week 16
Change in Health-related quality of life (HRQoL, measured by KCCQ-12) from baseline to week 16 | baseline to week 16
  KCCQ = Kansas City Cardiomyopathy Questionnaire
  The KCCQ 12 is a health-related quality of life questionnaire to measure the disease-specific health status of patients with heart failure. It is a 12 item questionnaire that quantifies physical function, symptoms (frequency, severity and recent change), social function, self-efficacy and knowledge and quality of life. Scores are generated for each domain and scaled from 0 to 100, with 0 denoting the lowest reportable health status and 100 the highest reportable health status.
Change in serum N-terminal pro brain natriuretic peptide (NT-proBNP) from baseline to week 16 | baseline to week 16
Change in echocardiographic markers of left ventricular function from baseline to week 16 | baseline to week 16
  measurement of left ventricular ejection fraction
Change in echocardiographic markers of left ventricular function from baseline to week 16 | baseline to week 16
  measurement of left ventricular diameter
Change in echocardiographic markers of left ventricular function from baseline to week 16 | baseline to week 16
  measurement of left ventricular end-systolic volume index
Change in echocardiographic markers of left ventricular function from baseline to week 16 | baseline to week 16
  measurement of left ventricular end-diastolic volume index
Change in echocardiographic markers of left ventricular function from baseline to week 16 | baseline to week 16
  measurement of left ventricular wall thickness
Change in echocardiographic markers of left ventricular function from baseline to week 16 | baseline to week 16
  measurement of left atrial volume index
Change in echocardiographic markers of left ventricular function from baseline to week 16 | baseline to week 16
  measurement of global longitudinal strain
Change in echocardiographic marker of left ventricular function from baseline to week 16 | baseline to week 16
  measurement of marker of diastolic function (E/e')
Change in echocardiographic markers of right ventricular function from baseline to week 16 | baseline to week 16
  measurement of right ventricular diameter
Change in echocardiographic markers of right ventricular function from baseline to week 16 | baseline to week 16
  measurement of tricuspid annular plane systolic excursion
Change in echocardiographic markers of right ventricular function from baseline to week 16 | baseline to week 16
  measurement of estimated systolic pulmonary arterial pressure
Liver: Change in Albumin from baseline to week 16 | baseline to week 16
Liver: Change in Alanine transaminase (ALT) from baseline to week 16 | baseline to week 16
Liver: Change in Aspartate transaminase (AST) from baseline to week 16 | baseline to week 16
Liver: Change in Bilirubin from baseline to week 16 | baseline to week 16
Kidney: Change in Creatinine (+Glomerular filtration rate) from baseline to week 16 | baseline to week 16
Change in New York Heart Association (NYHA) class from baseline to week 16 | baseline to week 16

OTHER OUTCOMES:
Incidence of treatment-emergent adverse events (AEs) | up to Week 20
  To assess the safety and tolerability of oral ferric maltol in heart failure patients with iron deficiency and anaemia.
Incidence of Adverse Events | up to Week 20
  Number of drop-outs due to AEs

CONTACTS AND LOCATIONS:
Overall Officials: Johann Bauersachs, Prof. Dr., Principal Investigator — Hannover Medical School, Department of Cardiology and Angiology
Locations (1):
- Hannover Medical School, Department of Cardiology and Angiology, Hanover, Lower Saxony, Germany

IPD SHARING:
Plan to Share IPD: No